CLINICAL TRIAL: NCT03516526
Title: Towards Personalized Dosing of Natalizumab in Multiple Sclerosis
Acronym: PDNMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Prothya Biosolutions (Industry); Erasmus Medical Center (Other); St. Antonius Hospital (Other); OLVG (Network); Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Zoé van Kempen, Coordinating investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL56584.029.16
Record Dates: First submitted 2018-04-12; First posted 2018-05-04 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Multiple Sclerosis
Keywords: natalizumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients in this study (Other): Patients treated with natalizumab with a minimum of 1 year, without signs of disease activity (relapses, new T2 lesions on MRI) for a minimum of 1 year.
  Interventions: Drug: Natalizumab

INTERVENTIONS:
Drug: Natalizumab — Extending dose intervals of natalizumab from 4 weeks to maximum of 8 weeks based on trough natalizumab concentrations

SUMMARY:
A prospective clinical trial with the aim of maintaining drug efficacy of natalizumab while extending dose intervals guided by drug concentrations in patients with relapsing remitting multiple sclerosis.

DETAILED DESCRIPTION:
Our main objective is to prove that extending dose intervals guided by natalizumab serum concentrations, will not result in radiological or clinical disease activity in completely stable RRMS patients treated with natalizumab. Adult patients with RRMS with no evident disease activity during the last 12 months of natalizumab infusions with a minimum treatment of 12 months wil be included. Before subsequent natalizumab infusions, serum concentrations will be evaluated. If the concentration exceeds 15μg/ml the dose interval will be extended with a week to a maximum of eight weeks. Patients will get regular brain MRI scans and clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing-remitting multiple sclerosis (RRMS) according to the McDonald criteria, revised by Polman 2010
* Natalizumab treatment for 12 months or longer at inclusion.
* An expanded disability status scale (EDSS) score of 0.0-6.0 at baseline.
* Natalizumab level of ≥15 μg/ml
* Written informed consent.

Exclusion Criteria:

* Any MS disease activity (radiologically or clinically) during the last 12 months of natalizumab treatment.
* Unable to undergo frequent MRI.
* The use of other immunomodulatory medication other than natalizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Gadolinium enhancing T1 lesions on brain MRI | 12 months
  Occurrence and number of gadolinium enhancing T1 lesions of brain MRI

SECONDARY OUTCOMES:
New T2 lesions on brain MRI | 12 months
  Occurrence and number of new T2 lesions on brain MRI
Relapses | 12 months
  scoring MS exacerbations
EDSS | 12 months
  Expanded Disability Status Scale: clinical scoring of disability in MS patients
MSFC | baseline and 12 months
  Multiple Status Functional Composite: clinical scoring of disability in MS patients
patient perspective measured with the SF-36 | baseline and 12 months
  questionnaire: Short Form-36
patient perspective measured with the MSIS-29 | baseline and 12 months
  questionnaire: Multiple Sclerosis Impact Scale-29

CONTACTS AND LOCATIONS:
Overall Officials: Joep Killestein, Dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (5):
- Netherlands (5):
  - OLVG, Amsterdam
  - VU medical center, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Erasmus medical center, Rotterdam
  - St. Antonius Hospital, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided